CLINICAL TRIAL: NCT03153592
Title: Effects of Mechanical Ventilation Guided by Transpulmonary Pressure on Gas Exchange During Robotic Surgery
Brief Title: Effects of Mechanical Ventilation Guided by Transpulmonary Pressure on Gas Exchange During Robotic Surgery: a Pilot Study
Acronym: Vetrapo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Gianmaria Cammarota, Physician in staff of the ICU, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CE 62/17
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Artificial Respiration; Surgery; Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will not know the arm of assignment. Care providers and investigators will know the arm, making the masking not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional ventilation strategy (Active Comparator): 13 patients will undergo volume controlled ventilation set with a tidal volume between 6-8 ml/kg of ideal body weight, positive end-expiratory pressure and fraction of inspired oxygen set to obtain a peripheral saturation in oxygen equal or greater than 94% and a plateau pressure <28 cmH2O.
  Interventions: Procedure: Conventional ventilation strategy
- transpulmonary pressure strategy (Experimental): 13 patients will undergo volume controlled ventilation set with a tidal volume at 6-8 ml/kg of ideal body weight, and with a inspiratory transpulmonary pressure less than 20 cmH2O and an expiratory transpulmonary pressure and inspired oxygen set accordingly to predefined criteria.
  Interventions: Procedure: Transpulmonary pressure driven ventilation strategy

INTERVENTIONS:
Procedure: Transpulmonary pressure driven ventilation strategy — Patients will receive volume controlled ventilation set with a tidal volume at 6-8 ml/kg of ideal body weight, an inspiratory transpulmonary pressure less than 20 cmH2O, and an expiratory transpulmonary pressure (PLexp) equal or greater than 0. At PLexp increasing from 0 up to 10 cmH2O, inspired fraction of oxygen would also be increased from 40% to 100%. Respiratory rate will be set to obtain an arterial partial pressure of carbon dioxide between 35 and 45 mmHg and to ensure a physiological pH. Whenever the clinician will deem it appropriate, an alveolar recruitment maneuver as previously described
  Arms: transpulmonary pressure strategy
Procedure: Conventional ventilation strategy — 13 patients will undergo volume controlled ventilation set with a tidal volume between 6-8 ml/kg of ideal body weight, positive end-expiratory pressure and fraction of inspired oxygen set to obtain a peripheral saturation in oxygen equal or greater than 94% and a plateau pressure <28 cmH2O Respiratory rate will be set to obtain an arterial partial pressure of carbon dioxide between 35 and 45 mmHg and in any case to ensure a physiological pH. In addition, whenever the clinician will deem it appropriate, an alveolar recruitment maneuver will be performed as previously described
  Arms: conventional ventilation strategy

SUMMARY:
Laparoscopy and robotic techniques are widespread procedures for pelvic gynecologic, urologic and abdominal surgery often performed in Trendelenburg position, with the application of pneumoperitoneum by inflating carbon dioxide. The rise in abdominal pressure following pneumoperitoneum and the head down body position have been shown to impair the respiratory function during the procedure, mainly inducing atelectasis formation in the dependent lung regions, worsening stress and strain of the alveolar structure.

The application of a ventilator strategy providing positive end-expiratory pressure (PEEP) has been shown to reduce the diaphragm cranial shift, increasing functional residual capacity and decreasing respiratory system elastance. Furthermore, the application of recruiting maneuver followed by the subsequent application of PEEP improved oxygenation. These results are in accordance with finding by Talmor et al, evaluating the effect of a mechanical ventilation guided by esophageal pressure in acute lung injury patients.

However a comparison between an esophageal pressure piloted mechanical ventilation and a conventional low tidal ventilator strategy with adjunct of PEEP and recruitment maneuvers according to clinical judgment has never been investigated in patients undergoing robotic gynecologic, abdominal or urologic surgery. The investigators aim to compare the conventional ventilation strategy (i.e. with application of PEEP and recruitment manoeuvre) with a ventilation driven by transpulmonary pressure assessed through an esophageal catheter, in patients undergoing to robotic surgery, with respect to oxygenation, expressed in terms of arterial oxygen tension - inspired oxygen fraction ratio (PaO2/FiO2) (primary endpoint), intraoperative respiratory mechanics indexes, number of lung recruitment maneuvers, rate and type of perioperative complications until hospital discharge (additional endpoint).

DETAILED DESCRIPTION:
INTRODUCTION Laparoscopy and robotic techniques are widespread procedures for pelvic gynecologic, urologic and abdominal surgery often performed in Trendelenburg position. Furthermore, in order to ameliorate surgical procedures, pneumoperitoneum is applied by inflating carbon dioxide. However, the rise in abdominal pressure following pneumoperitoneum and the head down body position have been shown to impair the respiratory function during the procedure, mainly inducing atelectasis formation in the declive lung regions. Consequently, functional residual capacity decreases and the risk of perioperative complications, such as hypoxaemia, rises up, particularly if patients are obese. Formation of atelectasis may worsen stress and strain of the alveolar structure. Stress, strain and atelectrauma give rise to ventilator-induced lung injury.

Although the role of ventilator-induced lung injury during general anesthesia is unclear, several investigations have been conducted with the purpose of improving arterial oxygenation and respiratory mechanics during laparoscopy. A ventilator strategy providing positive end-expiratory pressure (PEEP) has been shown to reduce the diaphragm cranial shift, increasing functional residual capacity and decreasing respiratory system elastance, principally in the obese subjects. Furthermore, the application of recruiting maneuver followed by the subsequent application of PEEP improved oxygenation during laparoscopy. Cinnella et al. demonstrated that an open lung strategy, i.e. a ventilation supported by recruiting maneuvers followed by the subsequent application of PEEP applied after pneumoperitoneum induction, increased transpulmonary pressure and led to alveolar recruitment and improvement of elastance of chest wall and gas exchange. These results are in accordance with finding by Talmor et al, evaluating the effect of a mechanical ventilation guided by esophageal pressure in acute lung injury patients.

However a comparison between an esophageal pressure piloted mechanical ventilation and a conventional low tidal ventilator strategy with adjunct of PEEP and recruitment maneuvers according to clinical judgment has never been investigated in patients undergoing robotic gynecologic, abdominal or urologic surgery.

Aim The investigators aim to compare the conventional ventilation strategy (i.e., with application of PEEP and recruitment manoeuvre) with a ventilation driven by transpulmonary pressure assessed through an esophageal catheter, in patients undergoing to robotic surgery, with respect to oxygenation, expressed in terms of arterial oxygen tension - inspired oxygen fraction ratio (PaO2/FiO2) (primary endpoint), intraoperative respiratory mechanics indexes, number of lung recruitment maneuvers, rate and type of perioperative complications until hospital discharge (additional endpoint).

METHODS Patients For this protocol, after informed consent has been obtained, 26 patients will be enrolled in the pilot randomized interventional study, eligible for robotic gynecological, urological and abdominal surgery at Maggiore Hospital Novara Italy.

1. The inclusion criteria will be: minimum age 18 years old, ASA I-II.
2. The exclusion criteria are: pre-existing lung and cardiac conditions that may lead to asa> II, contraindications to the positioning of a naso-gastric tube.

Intervention After the induction of general anesthesia, a naso-gastric tube equipped with gastric and esophageal balloon will be inserted (Nutrivent® - Seda). The nasogastric tube will be positioned and the esophageal balloon will be calibrated according to the findings by Mojoli et al.

In this phase, all patients will be ventilated a tidal volume (VT) of 6-8 ml / kg, in a volume controlled mode; PEEP (positive end-expiratory pressure) equal to zero and FiO2 set to obtain peripheral oxygen saturation (SpO2) > or = to 94% . The respiratory rate will be set to obtain arterial carbon dioxide tension (PaCO2) values between 35 and 45 mmHg and to ensure a physiological pH. At most, both a mild hypercapnia and a mild acidosis will be allowed.

In all the patients radial artery will be cannulated to monitor continuous intra-arterial blood pressure as usual practice, after Allen test results positive. The invasive hemodynamic monitoring will be performed through MOSTCARETM technology.

Subsequently, pneumoperitoneum will be applied to the patients, and the final position on the surgical table will be guaranteed. At this point, a recruitment maneuver will be applied, i.e., the ventilator is switched to pressure control ventilation, inspiratory time is increased to 50%, the peak inspiratory pressure gradient (above PEEP) is set at 20 cm H2O, and PEEP is progressively increased to obtain a stepwise increase of peak inspiratory to 30, 35, and 40 cm H2O every three breaths. The final recruiting pressure of 40 cm H2O is applied for six breaths. after recruiting maneuver ventilator is switched to previous ventilation mode. This maneuver is normally used to distend the lungs and prevent atelectasis .

Then, patients will be randomized into two groups according to a randomization list generated by a dedicated software. Clinician, at the surgical table, will open a sequentially numbered, opaque, sealed envelope to allocate the patient according to the randomization group. A researcher, not involved in the clinical care of the patient, will keep the randomization list. Patients will be randomized into:

1. Control group: 13 ventilated patients in Volume controlled VT 6-8 ml / kg; PEEP, and Fio2 (fraction of inspired oxygen) set for SpO2> or = to 94%, Plateau pressure <28 cm H2O.
2. Case group: 13 ventilated patients with current volume VT 6-8 ml / kg and in any case with a transpulmonary inspiratory pressure (PLinsp) of less than 20 cmH2O and transpulmonary expiratory pressure (PLexp) - FiO2, according to predefined criteria.

In both groups the respiratory rate will be set to obtain PaCO2 values between 35 and 45 mmHg and in any case to ensure a physiological pH. In addition, whenever the clinician will deem it appropriate, an alveolar recruitment maneuver will be applied, as previously described, in order to improve the PaO2 / FiO2 relationship.

Safety criteria In the intervention group in case of SpO2< to 94%, alveolar recruitment maneuvers will be applied.

Measurements During the study the following parameters will be recorded: arterial blood gas, respiratory mechanics parameters (airway pressure, tidal volume, transpulmonary pressure, flow, esophageal pressure),peritoneal insufflation pressure.

These measurement will be will be performed at:

1) 15 min after induction of anesthesia (STEP 1) 2) immediately after the positioning of the patient and / or the pneumoperitoneum induction (STEP 2) 3) immediately after the recruitment maneuver (STEP 3) 4) 20 minutes after the application of the ventilatory strategy select with the randomization (STEP 4) 5) after 60 minutes from the application of the ventilatory strategy select with the randomization (STEP 5) 7) every 60 minutes from the last step (STEP 6) 8) at the end of surgery after the elimination of the pneumo-peritoneum and / or in the supine position (STEP 7).

9) 1h after recovery from anesthesia (STEP 8). With the patient awake (i.e.before and after surgery), a lung ultrasound will be carried out to evaluate the degree of ventilation / atelectasis .

Statistical analysis For this pilot randomized study, was calculated a sample size of 26 patients in total i.e., 13 patients per arm . To determine sample size, the investigators expected a difference of 80 mmHg between the mean value of PaO2/FiO2 of the two groups and a standard deviation of 60 mmHg, with a power of 80% and an alpha of 0.05.

The continuous variables will be presented as the median and interquartile and will be compared using the Mann Whitney test. Categorical variables, whether dichotomous or nominal, will be evaluated with a Fisher test. A trend analysis will be carried out within each group over the course of each step.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score I - II
* Patients requiring elective robotic gynecological-abdominal surgery

Exclusion Criteria:

- Contraindications to the positioning of a naso-gastric tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Oxygenation Changes | Soon after anesthesia induction (step 1), after 45 min from step 1 (pneumoperitoneum, trendelemburg, recruitment maneuver application-step 2),after 20min from randomization (step 3), every 60 min during surgery and at its end, after 1 hour from recovery.
  Ratio between the arterial partial pressure (PaO2) and inspired fraction (FiO2) of oxygen (PaO2/FiO2)

SECONDARY OUTCOMES:
Intraoperative respiratory mechanics indexes changes | Soon after anesthesia induction (step 1), after 45 min from step 1 (pneumoperitoneum, trendelemburg, recruitment maneuver application-step 2),after 20min from randomization (step 3), every 60 min during surgery and at its end, after 1 hour from recovery.
  Airway pressure, flow, esophageal and transpulmonary pressures
Number of lung recruitment maneuvers | During the whole surgical procedure
  The number of recruitment maneuvers required during the surgery will be recorded
Type of perioperative complications | within the following 30 days after surgery
  postoperative hypoxemia, presence of lung atelectasis, occurrence of pneumonia, sepsis, severe sepsis or septic shock
Rate of perioperative complications | within the following 30 days after surgery
  Number of perioperative complication occurred during the hospital length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Maggiore della Carita, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valenza F, Chevallard G, Fossali T, Salice V, Pizzocri M, Gattinoni L. Management of mechanical ventilation during laparoscopic surgery. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):227-41. doi: 10.1016/j.bpa.2010.02.002. PMID 20608559
- [Background] Strang CM, Hachenberg T, Freden F, Hedenstierna G. Development of atelectasis and arterial to end-tidal PCO2-difference in a porcine model of pneumoperitoneum. Br J Anaesth. 2009 Aug;103(2):298-303. doi: 10.1093/bja/aep102. Epub 2009 May 13. PMID 19443420
- [Background] Perilli V, Sollazzi L, Bozza P, Modesti C, Chierichini A, Tacchino RM, Ranieri R. The effects of the reverse trendelenburg position on respiratory mechanics and blood gases in morbidly obese patients during bariatric surgery. Anesth Analg. 2000 Dec;91(6):1520-5. doi: 10.1097/00000539-200012000-00041. PMID 11094011
- [Background] Chiumello D, Carlesso E, Cadringher P, Caironi P, Valenza F, Polli F, Tallarini F, Cozzi P, Cressoni M, Colombo A, Marini JJ, Gattinoni L. Lung stress and strain during mechanical ventilation for acute respiratory distress syndrome. Am J Respir Crit Care Med. 2008 Aug 15;178(4):346-55. doi: 10.1164/rccm.200710-1589OC. Epub 2008 May 1. PMID 18451319
- [Background] Pelosi P, Ravagnan I, Giurati G, Panigada M, Bottino N, Tredici S, Eccher G, Gattinoni L. Positive end-expiratory pressure improves respiratory function in obese but not in normal subjects during anesthesia and paralysis. Anesthesiology. 1999 Nov;91(5):1221-31. doi: 10.1097/00000542-199911000-00011. PMID 10551570
- [Background] Futier E, Constantin JM, Pelosi P, Chanques G, Kwiatkoskwi F, Jaber S, Bazin JE. Intraoperative recruitment maneuver reverses detrimental pneumoperitoneum-induced respiratory effects in healthy weight and obese patients undergoing laparoscopy. Anesthesiology. 2010 Dec;113(6):1310-9. doi: 10.1097/ALN.0b013e3181fc640a. PMID 21068660
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Derived] Cammarota G, Lauro G, Sguazzotti I, Mariano I, Perucca R, Messina A, Zanoni M, Garofalo E, Bruni A, Della Corte F, Navalesi P, Bignami E, Vaschetto R, Mojoli F. Esophageal Pressure Versus Gas Exchange to Set PEEP During Intraoperative Ventilation. Respir Care. 2020 May;65(5):625-635. doi: 10.4187/respcare.07238. PMID 32345760